CLINICAL TRIAL: NCT01503528
Title: Outcomes After Total Knee Joint Arthroplasty: A Comparative Study Using 3 Different Analgesic Techniques
Brief Title: Motor Sparing Block vs. Peri-Articular Catheters
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Shortage of required study drug.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, James Howard, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18448; 101754 (Other: Research and ethics board, University of Western Ontario)
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Knee Joint Arthritis; Knee Joint Arthroplasty
Keywords: arthroplasty; wound; catheter; local; anesthesia; infiltration; Total Knee Arthroplasty
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized clinical trial. For safety and logistical reasons, it cannot be blinded. In the perioperative period multiple factors contribute to discharge readiness. The major impediments to early discharge include poor pain control, opioid related adverse events, surgical/ medical complications, inability to achieve physiotherapy end points and patient's unwillingness to be discharged. We want to compare head to head, two previously evaluated fast-track paradigms. We are not comparing just the analgesic technique alone. We are comparing the pathways where the analgesic regimes are a component and differ, keeping the common factors similar between the groups. If a technique does not allow early ambulation, patients cannot be ready for discharge and thus resource utilization will be affected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Sparing Nerve Block (Active Comparator): Motor sparing knee block (60mL of 0.5% ropivacaine with 10 mg Morphine, 30 mg Ketorolac and 150 mcg of epinephrine as the initial bolus) initiated in the preoperative period in the block room as per the standard practice and continued until discharge. Spinal anesthetic with 15 mg of hyperbaric bupivacaine. Patients will be connected to an Ambit infusion pump in the postoperative period set to deliver ropivacaine 0.2% at a basal infusion rate of 7 mL/Hr with patient controlled boluses of 5mL every hour for breakthrough pain. Patients will be discharged home following removal of the anaesthetic catheter and fulfilling criteria for discharge.
  Interventions: Procedure: Motor Sparing Nerve Block
- Peri-Articular Catheters (Experimental): 3 peri-articular catheters inserted at the end of surgery followed by peri-articular infiltration with ropivacaine 0.2% and wound infusions will be continued until discharge using elastomeric devices. Spinal anesthetic with 15 mg of hyperbaric bupivacaine. Patients will be discharged home following removal of the anaesthetic catheter and fulfilling criteria for discharge.
  Interventions: Procedure: Peri-articular Catheters

INTERVENTIONS:
Procedure: Motor Sparing Nerve Block — Continuous Motor sparing knee block (60mL of 0.5% ropivacaine with 10 mg Morphine, 30 mg Ketorolac and 150 mcg of epinephrine as the initial bolus) initiated in the preoperative period in the block room as per the standard practice and continued until discharge. Patients will be connected to an Ambit infusion pump in the postoperative period set to deliver ropivacaine 0.2% at a basal infusion rate of 7 mL/Hr with patient controlled boluses of 5mL every hour for breakthrough pain.
  Arms: Motor Sparing Nerve Block
Procedure: Peri-articular Catheters — 3 peri-articular catheters inserted at the end of surgery followed by periarticular infiltration with ropivacaine 0.2% and wound infusions will be continued until discharge using elastomeric devices.
  Arms: Peri-Articular Catheters

SUMMARY:
This study is designed to determine if one anaesthetic modality, either motor sparing nerve block or peri-articular local infiltration anaesthesia with infusion, is superior in providing postoperative analgesia following total knee joint arthroplasty and if the efficacy of analgesia affects TKA outcomes. These outcomes include pain and function for a period of up to 3 months, narcotic consumption, and specific non-pain complications, including cardiac, respiratory, central nervous system, thromboembolism, infection, nausea and vomiting and urinary retention.

Economic outcomes will also be examined, including length of hospital stay, direct health care costs and patient satisfaction.

DETAILED DESCRIPTION:
Seventy patients of either sex with ASA physical status of 1-3, aged greater than 30 years scheduled for elective primary unilateral total knee arthroplasty will be the randomized to one of 2 groups. The patients will be identified by the surgeons and seen in the pre-admit clinic to obtain informed consent, and collect health and joint related data using SF-12, Knee Society Scores, and WOMAC surveys. The randomization will occur in the pre-admit clinic with a closed envelope system. This is not a blinded study for logistical reasons.

Group 1: Control- Motor Sparing Nerve Block Continuous Motor sparing knee block (using 60mL of 0.5% Ropivacaine with 10 mg Morphine, 30 mg Ketorolac and 150 mcg of epinephrine as the initial bolus) initiated in the preoperative period in the block room by anesthesia as per the standard practice( 25mL for posterior knee infiltration, 5mL for LFCN, 25mL for adductor canal under the fasica lata, 5ML for intermediate cutaneous nerve of thigh) and continued until discharge. CADD infusion pump will deliver Ropivacaine 0.2% at a basal infusion rate of 8 mL/Hr with no patient controlled boluses.

Group 2: Intervention- Local Infiltration + Infusion Anesthetic Wound infiltration will first be completed per standard practice using 110mL of ropivacaine 300mg, ketorolc 30mg ,morphine 10mg for infiltration. After, three peri-articular catheters (inserted into the suprapatellar pouch, anterior subcutaneous cutaneous tissue, posterior to the femur) will be inserted at the end of the case followed by periarticular infusion with CADD infusion pump delivering Ropivacaine 0.2% at a basal infusion rate of 8 mL/Hr with no patient controlled boluses

All patients will receive sedation with fentanyl and midazolam titrated to effect during the initiation of spinals and MSNB blocks. All patients will receive intravenous sedation with an infusion of a mixture of propofol and ketamine titrated to effect during surgery. Patients will be discharged home following removal of the anaesthetic catheters and fulfilling criteria for discharge

All patients will receive standard multimodal analgesia pre- and post-operatively.

Pain scores, nausea/sedation, narcotic consumption, and any post-operative complications will be assessed and documented 6 hours post-op on the day of surgery. After this, pain scores will be documented twice daily till the end of pian study period (post-discharge day 4 and once more at 2 weeks post-op) and will be recored when at rest and with mobility (two VAS scores each assessment) . Nausea and sedation will be documented at time of assessment from the patient or nursing charts as well as the patient pain diary.

The discharge criteria is as follows

1. The patient should be able to take care of personal care, get in and out of bed, into and up from a chair, on and off a toilet and to walk with proper walking aids 70 m without time limit; ability to do five steps.
2. Free of medical or surgical complications including urinary catheterization or need for blood transfusion
3. Acceptable pain relief (NRS = 5/10) without any need for intravenous analgesics.
4. No nausea/ vomiting; generalized weakness or dizziness.
5. Knee flexion of 90 degreeed is optional but preferred.

The patients will be assessed at 6 hours of arrival to PACU and at 9 AM and 2pm on POD 1. If the patients were not discharged on POD 1 , the readiness for discharge will be at 9 AM on postoperative day 2 subsequently. WOMAC scores, KSS scores and SF-12 will be collected at the Pre-admit clinic and will be repeated at 6 weeks and three months postoperatively. Block performance characteristics prospectively collected will include procedural time, success, number of attempts and complications such as persistent paresthesia and intravascular injection. Inpatient assessment by the research team as well as a pain diary for documentation following discharge will be used to collect data including numeric pain score on movement and rest at various time intervals (twice daily), the predominant site of pain, frequency of rescue analgesic consumption, total analgesic consumption, symptoms of sedation and nausea for up to 4 days post-discharge. Time to first physiotherapy session and their progress/ability to perform rehabilitation exercises daily will be documented. Regardless of the group the patient is randomized to, their anesthetic device (MSNB or LIA infusion) will be discontinued and removed in hospital prior to discharge. Time to discharge readiness and actual duration of hospital stay will be documented.

Total patient involvement time is 3 months (from surgery to 3 month follow-up appointment).

In hospital, adverse events will be retrieved from patient charts and nursing/physician documentation. Post discharge adverse events will be collected by the patient diary and at their 2 weeks, 6 week and 3 month post-operative follow-up. These will include occurrence of myocardial events, DVT, Pulmonary emboli, delirium, pneumonia, paralytic ileus, gastrointestinal bleed, new onset renal dysfunction and wound infection.

Delayed or post- discharge adverse events and duration of narcotic therapy will be collected in the out-patient clinic at 2 weeks and at 6 weeks and 3 months after surgery at their follow-up appointment.

Wound and prosthetic infections and the presence of chronic post-surgical pain will be recorded from the surgical follow up notes.

Primary hypothesis (null):

The post-operative inpatient stay and discharge rates following TKJA are comparable between motor sparing knee blocks and peri-articular wound catheters.

Secondary hypotheses (null):

1. Pain scores and analgesic consumption with motor sparing block or by peri-articular wound catheters are comparable.
2. Adverse events and complication rates are comparable between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Adult patients ASA physical status 1-3, Ability to give informed consent, No contraindications to regional techniques, Ability to perform study related tests, Scheduled for primary unilateral total knee arthroplasty

Exclusion Criteria:

Revision of arthroplasty, Allergy to local anesthetics and multimodal analgesic drugs, Contraindications to spinal anesthesia, Inability to perform study related procedures, Inability to give informed consent, Wheel chair bound, Pregnancy, Chronic renal failure, BMI >45

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome - Perioperative pain | day of surgery to 2 weeks post-op
  Postoperative pain levels on a visual analogue scale will be recorded while the patient is an inpatient up to a maximum of 4 days post-discharge, and again at 2 weeks post-op.

SECONDARY OUTCOMES:
Readiness and True Discharge times | in-patient period
  Readiness for discharge and the actual time of discharge will be recorded
Postoperative mobility/function | Measured on day of surgery to discharge day 4. Functional outcomes will be collected at 6 weeks and 3 months post-op using WOMAC and KSS scores
  Postoperative mobility will be assessed by a physiotherapist, and recorded using inpatient assessment notes and patient recorded physiotherapy progression following discharge in their pain diary.
Analgesia/Narcotic Consumption | day of surgery to post-discharge day 4
  Break-through/rescue analgesia and narcotics that were consumed between assessment intervals will be documented
Complications | day of surgery to 3 months post-op
  Post-operative complications such as myocardial events, DVT, Pulmonary emboli, delirium, pneumonia, paralytic ileus, gastrointestinal bleed, new onset renal dysfunction and wound infection
Nausea and Sedation symptoms | day of surgery to post-discharge day 4
  Analgesic side-effects will be monitored and compared to narcotic consumption
Patient reported pain, stiffness and functional disability. | Assessed preoperatively, and at 6 weeks and 3 months postoperative.
  These variables will be assesed using the Knee Society Score and Western Ontario and McMaster Universities Arthritis Index (WOMAC score).
Short-From Survey-12 | Assessed preoperatively, and at 6 weeks and 3 months postoperative.
  Overall assessment of patient's health
Anaesthetic Procedure Performance Data | peri-operatively
  Block performance characteristics prospectively collected will include procedural time, success, number of attempts and complications such as persistent paresthesia and intravascular injection

CONTACTS AND LOCATIONS:
Overall Officials: James Howard, FRCSC, Principal Investigator — Associate Professor, London Health Sciences Centre
Locations (1):
- London Health Sciences Centre University Hospital, London, Ontario, Canada